CLINICAL TRIAL: NCT06733103
Title: Adapted Cognitive Stimulation Therapy (CST) for Pre-frail Stroke Survivors: A Non-randomised, Acceptability and Feasibility Pilot Study
Brief Title: Pilot of Cognitive Stimulation Therapy for Pre-frail Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 335493
Record Dates: First submitted 2024-12-03; First posted 2024-12-13 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Frailty; Carers
Keywords: FIESTO; sCST
MeSH Terms: conditions — Stroke; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sCST Intervention Group (Experimental): There is only one arm of this intervention, it involves stroke survivors attending a cognitive stimulation group designed for post-stroke frailty. This involves strategies and psychoeducation and take-home sheets for stroke survivors and their carers. After the group is finished, stroke survivors will attend interviews and the findings of these interviews will be analysed through the theoretical framework of accepatability. The same will be the case for carers.
  Interventions: Behavioral: Stroke Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Stroke Cognitive Behavioural Therapy — This is the only intervention in this clinical (feasibility) study

SUMMARY:
Frailty is described as a type of vulnerability where one can struggle to recover fully from things that can put stress on one's body, e.g., cold weather or bronchitis. This can lead to negative health outcomes and is linked with early death, particularly if the person has had a stroke. Frailty was first operationalised by Fried et al. (2001) as the presence of at least three out of the following five clinical indicators: unintentional weight loss, exhaustion, weakness, slow walking speed and low level of physical activity. They also defined 'intermediate frailty status', now referred to as 'pre-frailty', as the occurrence of one or two of the five criteria.

An alternative perspective on frailty was proposed by Mitnitski et al. (2001), suggesting it refers to the number of health deficits an individual has accumulated. Individuals assessed as pre-frail have an increased risk of becoming frail in the following few years, and those assessed as frail are more likely to die (Gill et al., 2006). However, frailty is potentially reversible at the pre-frail stage, making pre-frailty an important target for intervention (Gill et al., 2006).

A promising approach to the reversal of pre-frailty is multicomponent interventions consisting of a physical exercise intervention combined with nutritional, cognitive, social and/or other interventions, which have been shown to reduce frailty ratings in pre-frail older adults (aged 65 or above) (Apóstolo et al., 2018; Dedeyne et al., 2017; Tam et al., 2022).

Interestingly, cognitive training interventions alone can also have a positive impact on frailty ratings (Ng et al., 2015), indicating a potential role for psychologically informed interventions in frailty management. If multicomponent interventions reverse frailty in pre-frail older adult populations, it is possible they may also reverse frailty in pre-frail stroke populations and help to reduce the risk of associated adverse outcomes.

There is limited consistency across the existing literature of multicomponent interventions regarding the mode of delivery, content, and duration of the cognitive component (e.g. Apóstolo et al., 2019; Chen et al., 2020; Murukesu et al., 2020; Ng et al., 2015). However, some formats of the cognitive interventions used share similarities with Cognitive Stimulation Therapy (CST; Spector et al., 2003). CST is an intervention for individuals with mild to moderate dementia and is recommended by the National Institute of Health and Care Excellence [NICE] (2018); it has been researched globally and found to improve cognition, quality of life, well-being, mood and activities of daily living (Aguirre et al., 2013; Lobbia et al., 2019).

CST might, therefore, provide a good basis for the cognitive training component of a multicomponent frailty intervention, including within stroke populations. However, there is currently no research applying CST in a population where stroke is the primary diagnosis. We therefore want to find out if an adapted version of CST will be a feasible and acceptable intervention for stroke survivors and their informal carers, who have been found to spend over 30 hours per week supporting the stroke survivor (Deloitte Access Economics, 2020).

The thoughts of the stroke survivors (who will have attended the pilot group intervention) and their carers (who will have not attended the intervention but will have supported the stroke survivor to attend and complete between session activities) will be gathered from focus groups. We will explore their thoughts on the feasibility and acceptability of the intervention (fore example, whether it can be reasonably carried out and is felt to be appropriate).

This study is part of a larger research project on Frailty and its Effects on Stroke Treatments and Outcomes (FIESTO) and the findings will inform the neuropsychological component used in a feasibility randomised control trial investigating a multicomponent intervention for pre-frail stroke survivors.

DETAILED DESCRIPTION:
Purpose and Design Frailty is a state of vulnerability characterised by multi-system decline in physiological reserves needed to maintain homeostasis following a stressor e.g., cold weather or bronchitis (Morley et al., 2013; Fried et al., 2001; Campbell & Buchner, 1997). Fried et al (2001) operationalise frailty as the presence of three or more indicators in terms of shrinking (unintentional weight loss of 10 lbs or more in the last year), self-reported exhaustion, weakness of grip strength, slowness of walking speed, or low physical activity. Poorer functional outcomes such as higher rates of institutionalisation, and increased rates of mortality and illness are common (Wallis et al., 2015; Fried et al., 2001). Pre-frailty is the presence of one or two indicators and is associated with elevated risk of adverse outcomes and of declining into frailty (Fried et al., 2001). Gill et al. (2006) found people who were pre-frail were likely to transition to frailty, and people who were frail were three to five times more likely to die over the course of their 54-month study.

Importantly, however, they found frailty can be reversed with interventions delivered at the pre-frail stage (Fried et al., 2001; Ng et al., 2015; Gill et al., 2006).

Promising approaches to the reversal of pre-frailty and associated negative outcomes are multicomponent interventions that consist of a physical exercise intervention combined with nutritional, cognitive, social and/or other interventions. These have been shown to reduce frailty ratings in pre-frail older adults (aged 65 or above) (Apóstolo et al., 2018; Dedeyne et al., 2017; Tam et al., 2022). Interestingly, cognitive training interventions alone can also have a positive impact on frailty ratings (Ng et al., 2015), indicating a potential role for psychologically informed interventions in frailty management. Given multicomponent interventions can reverse frailty in pre-frail older adult populations, it is possible they may also reverse frailty in pre-frail stroke populations and help to reduce the risk of associated adverse outcomes.

Dr Nicholas Evans, Honorary Consultant in Stroke Medicine at Addenbrooke's Hospital and Senior Clinical Lecturer at the University of Cambridge, is leading the 'Frailty and Its Effects on Stroke Treatments and Outcomes' (FIESTO) project, supported by the Stroke Association. This will include a feasibility Randomised Controlled Trial (RCT) of a multicomponent intervention consisting of physical, cognitive and nutritional components for pre-frail stroke survivors in preparation for a full-scale RCT. However, initial work is required to develop each individual component of the overall multicomponent intervention.

There is limited consistency across the existing literature of multicomponent interventions regarding the mode of delivery, content, and duration of the cognitive training component (e.g. Apóstolo et al., 2019; Chen et al., 2020; Murukesu et al., 2020; Ng et al., 2015). However, some formats of cognitive training used in these interventions share similarities with Cognitive Stimulation Therapy (CST; Spector et al., 2003). CST is an intervention for individuals with mild to moderate dementia and is recommended by the National Institute of Health and Care Excellence [NICE] (2018); it has been researched globally and found to improve cognition, quality of life, well-being, mood and activities of daily living (Aguirre et al., 2013; Lobbia et al., 2019). CST might, therefore, provide a good basis for the cognitive training component of a multicomponent frailty intervention, including within stroke populations. However, there is currently no research applying CST in a population where stroke is the primary diagnosis.

Two doctoral thesis projects will investigate the feasibility and acceptability of adapting CST for pre-frail stroke survivors. Acceptability will be investigated with the survivors who experience the intervention and the informal carers who support them with attendance and with between-session activities. The two lead researchers of these related studies will work together to adapt the CST intervention and co-facilitate the sessions for stroke survivors, however, data collection and analysis will be conducted independently.

Recruitment Participants for this study will be ten dyads of adult pre-frail stroke survivors (PfSS) and their informal carers (ICs). It is planned to recruit PfSS under the care of the Addenbrookes Hospital stroke services (Acute Stroke Unit and Lewin Rehabilitation Unit), either just before they go back home, or shortly after they have returned home from hospital. PfSS within six months post-stroke will be recruited in line with recruitment criteria for the future FIESTO trial and within this chronological window due to the time-sensitive nature of pre-frailty and its progression to frailty (Gill et al., 2006). The manual for Cognitive Stimulation Therapy suggests a group size of between five and eight, however recruiting for ten aims to account for participant attrition (Spector et al., 2006).

PfSS will be identified by clinicians working in Addenbrooke's stroke services based on the inclusion and exclusion criteria. Clinical Frailty Scale scores (CFS; Rockwood et al., 2005) scores and Oxford Cognitive Screening (OCS; Demeyere et al., 2015) scores are collected routinely by these clinicians and these scores will be used to help determine eligibility. To be eligible for participation, stroke survivors will need to score between three and four on the CFS and show impairment in at least one domain on the OCS. Addenbrooke's Hospital stroke services clinicians will be fully briefed in the inclusion and exclusion criteria of the study by the research team in a letter to recruiters. Clinicians who identify a patient as being potentially eligible for participation will raise this during the Multidisciplinary Team (MDT) meetings within the Addenbrooke's stroke services and Dr Nicholas Evans (Honorary Consultant in Stroke Medicine and Principal Investigator from Cambridge University Hospitals NHS Trust) or Dr Huw Green (Principal Clinical Psychologist in Stroke, a member of the clinical team as well as the research team) will review the clinical notes. Should they agree that the dyad appears eligible, the original clinician will provide the dyad with a 'consent to contact' form and a research poster. The dyad then have three methods via which they can express their interest to hear more from researchers about the study: 1) they can follow the web address/QR code to a Microsoft Forms 'Interest registration' document where they can provide their contact details to researchers and state their preferences for contact, 2) they can email the researchers directly, 3) they can complete the physical 'consent to contact' form which asks for contact details and preferences. If a 'consent to contact' form is completed, the stroke survivor's copy will be uploaded to their electronic records by a member of the clinical team.

If the patient and their informal carer complete one of the above expression of interest methods, one of the research team members (Sophie Livsey, Max Bramley, Dr Nicholas Evans or Dr Huw Green) will either visit the patient and carer on the ward or, if the stroke survivor has been discahrged home, contact them via their preferred method in order to discuss the study more and provide the information sheet (by email or post, if at home).

If the dyad is still interested in participating, a further visit (either on the ward or at their home) will be arranged with at least one of the lead researchers (Sophie Livsey and/or Max Bramley), after a minimum of 24 hours, in order to answer any further questions and go through the informed consent process.

If the participant or their carer are found to lack capacity to provide their informed consent to participate they will be sensitively informed that they do not meet eligibility criteria. The same applies if either the participant or their carer are found to lack sufficient English language ability to be able to engage effectively in a focus group.

Inclusion/Exclusion

Inclusion Criteria PfSS:

Within 6 months post-stroke Discharged home, or due to be discharged home before the intervention is to begin Pre-frail (scoring three or four on the CFS) Demonstrating impairment in at least one cognitive domain, according to the routinely-administered Oxford Cognitive Screen (Demeyere et al., 2015) Aged 18+ Have an informal carer willing to participate alongside them Have good English language ability

Exclusion Criteria PfSS:

Those deemed by the stroke team as lacking capacity to consent to participate in research. This will be screened initially by stroke team and again by researchers prior to informed consent process Dementia diagnosis No access (or ability or support to access) Microsoft Teams Significant language difficulties (assessed via clinical judgement as likely to impact their ability to participate in the focus group)

Inclusion Criteria IC:

Are an IC for a PfSS who meets the above inclusion criteria Have good English language ability

Exclusion Criteria IC:

Live separately from the PfSS Are subject to an active safeguarding investigation Significant language difficulties (assessed via clinical judgement as likely to impact their ability to participate in the focus group)

Providing care to the PfSS participant in a professional capacity

Those deemed by the stroke team as lacking capacity to consent to participate in research. This will be screened initially by stroke team and again by researchers prior to informed consent process

Consent All participants will be provided with an information sheet and will be asked to provide full, informed consent before entering the study. Potential participants will be given a minimum of 24 hours to review the participant information sheet to consider whether they wish to participate before the informed consent process begins. Addenbrookes Hospital stroke services clinicians will be asked to suggest potential participants who are deemed to possess mental capacity to participate in the research, this will be assessed again by researchers prior to the informed consent process.

As part of the consent process, PfSS paticipants will be required to consent to the researchers accessing their medical records.

Risks, burdens and benefits It is possible that taking part in this research may cause distress, harm or burden to participants. Anticipated risks, such as burden of time commitment, fatigue or clashes with fellow participants, will be outlined in the PIS.

The intervention will be delivered in a suitable room on the Cambridge Biomedical Campus which will be assessed for risks. Dr Nicholas Evans will be present during intervention sessions, as a member of Addenbrooke's Hospital staff and Consultant in Stroke Medicine, should any health-related risk issues arise during the group.

Participants will be encouraged to speak up should they experience any harm or distress as a result of the study, at which point effort will be made to resolve or reduce issues (e.g., difficult group dynamics may benefit from alternative seating arrangements) but participants will also be reminded of their right to withdraw from the study.

Although participants may experience some benefits from participating in this study (such as improvements to their psychological well-being or day-to-day functioning), benefits are not guaranteed; participants will be informed of this.

Study participation will require PfSS participants to donate approximately 10 hours of their time, and IC participants approximately 2 hours In addition, not including travel time.

There will be a financial cost of travelling to and from Addenbrooke's. Dr Evans, as a member of Addenbrooke's Hospital clinical staff, has also agreed to provide documentation that will allow participants to receive discounted parking at the hospital for the intervention sessions.

Coercion Although Dr Nicholas Evans (Honorary Consultant in Stroke Medicine and CUH Principal Investigator) and Dr Huw Green (Clinical Psychologist in Neuropsychology) have agreed to be involved in approaching potential participants about the study and providing the Participant Information Sheets, the lead researchers will take responsibility for the informed consent process as these researchers are not part of the patient's clinical team. If Dr Evans or Dr Green are involved in informed consent, the participants may feel more obligated to take part.

Nevertheless, it will be made clear to potential participants that there will be no consequences to their treatment if they choose not to take part, not if they withdraw from the study at a later date.

PfSS participants will be informed that if the do wish to participate in the study, they will remain open to Dr Nicholas Evans or one of his Consultant colleagues for follow-up in clinic 6-months after the study is complete. This is to ensure that participants will be able to be reviewed and receive care should anything arise during the course of the study that may require medical attention. Access to continued follow-up by a Consultant could be seen as a benefit to taking part however this is not intended to be coercive, but instead a safety precaution.

Confidentiality Participants will also be informed of how their information and the data the provide will be used. Participants will be made aware that due to the group nature of the intervention and focus group, that some personal information (such as first names or a preferred nickname) will need to be shared with other participants. However, participants will be informed that it will be up to them what other personal information they choose to disclose during these group activities.

PfSS participants will be informed that their medical records will be accessed in order to obtain additional information about their demographics (e.g., age, ethnicity, etc.), their stroke (e.g., type, location, etc.) and their resulting difficulties (e.g.,frailty and cognitive screening scores). They will be informed that any data collected from their medical records or from the focus groups will not be tied to any identifiable information such as their name. Their data will instead be assigned to an anonymous participant identification code when stored by the researchers. Personal/contact information will only be used by researchers for the purpose of communication and will be destroyed after the last communication with participants is complete. Participants will be made aware that some direct quotations may be taken from the focus group transcripts and published in the final report, however every effort will be taken to ensure that the participant cannot be identified from the published quotes.

All data will be stored securely on the password-protected Microsoft OneDrive for Business, a secure online storage platform linked to UEA in line with the UEA Data Management Policy (2022). Any data collected for the study will be kept for will be stored securely on the UEA One Drive for Business with the project supervisor, Dr Catherine Ford, becoming custodian for the data, once the lead researchers have completed their course and are no longer enrolled at UEA. The data will be kept in this location for 10 years after the findings are published and will then be deleted. Participants will be informed how their data will be stored before consenting to the study in accordance with The Data Protection Act (2018).

All identifiable data will be stored separately from the anonymised data on the OneDrive.

As per NHS guidelines, participants will be informed confidentiality can be broken if it is felt the individual is likely to come to immediate significant harm or cause significant harm based on disclosures to researchers and PfSS participants will be required, as part of the consent form, to consent to their GP being informed of their involvement in the research study.

Debrief/Conflict of Interest A debrief letter will be sent to participants as per the procedure. This will detail how to contact the research team, should participants have questions. This will also reiterate our thanks for participating and how study results will be communicated at a later date, with plans for publication. The participant information sheet will also explain that any decision about participation in the study will not affect their care from AHST, be this declining to participate or withdrawing from the study.

References Aguirre, E., Woods, R. T., Spector, A., & Orrell, M. (2013). Cognitive stimulation for dementia: A systematic review of the evidence of effectiveness from randomised controlled trials. Ageing Research Reviews, 12(1), 253-262.

https://doi.org/10.1016/j.arr.2012.07.001

Apóstolo, J., Cooke, R., Bobrowicz-Campos, E., Santana, S., Marcucci, M., Cano, A., Vollenbroek-Hutten, M., Germini, F., D'Avanzo, B., Gwyther, H., & Holland, C. (2018). Effectiveness of interventions to prevent pre-frailty and frailty progression in older adults: A systematic review. JBI Database of Systematic Reviews and Implementation Reports,16(1), 140-232.

https://doi.org/10.11124/JBISRIR-2017-003382

Apóstolo, J., Dixe, M. D. A., Bobrowicz-Campos, E., Areosa, T., Santos-Rocha, R., Braúna, M., Ribeiro, J., Marques, I., Freitas, J., Almeida, M. de L., & Couto, F. (2019). Effectiveness of a combined intervention on psychological and physical capacities of frail older adults: A cluster randomized controlled trial. International Journal of Environmental Research and Public Health, 16(17).

https://doi.org/10.3390/ijerph16173125

Campbell, A. J., & Buchner, D. M. (1997). Unstable disability and the fluctuations of frailty. Age Aging, 26, 315-318. Chen, L. K., Hwang, A. C., Lee, W. J., Peng, L. N., Lin, M. H., Neil, D. L., Shih, S. F., Loh, C. H., & Chiou, S. T. (2020). Efficacy of multidomain interventions to improve physical frailty, depression and cognition: data from cluster randomized controlled trials. Journal of Cachexia, Sarcopenia and Muscle, 11(3), 650-662.

https://doi.org/10.1002/jcsm.12534

Dedeyne, L., Deschodt, M., Verschueren, S., Tournoy, J., & Gielen, E. (2017). Effects of multi-domain interventions in (pre)frail elderly on frailty, functional, and cognitive status: A systematic review. Clinical Interventions in Aging, 12, 873- 896. https://doi.org/10.2147/CIA.S130794

Demeyere, N., Riddoch, M. J., Slavkova, E. D., Bickerton, W.-L., & Humphreys, G. W. (2015). The Oxford Cognitive Screen (OCS): Validation of a Stroke-Specific Short Cognitive Screening Tool. Psychological Assessment.

https://doi.org/10.1037/pas0000082.supp

Fried, L. P., Tangen, C. M., Walston, J., Newman, A. B., Hirsch, C., Gottdiener, J., Seeman, T., Tracy, R., Kop, W. J., Burke, G., & McBurnie, M. A. (2001). Frailty in Adults: Evidence for a Phenotype. Journal of Gerontology: Medical Sciences, 56(3), 146-156.

Gill, T. M., Gahbauer, E. A., Allore, H. G., & Han, L. (2006). Transitions Between Frailty States Among Community-Living Older Persons. Archives of International Medicine, 166, 418-423.

https://jamanetwork.com/

Lobbia, A., Carbone, E., Faggian, S., Gardini, S., Piras, F., Spector, A., & Borella, E. (2019). The Efficacy of CognitiveStimulation Therapy (CST) for People with Mild-to-Moderate Dementia: A Review. European Psychologist, 24(3), 257-277. https://doi.org/10.1027/1016-9040/a000342

Morley, J. E., Vellas, B., van Kan, G. A., Anker, S. D., Bauer, J. M., Bernabei, R., Cesari, M., Chumlea, W. C., Doehner, W., Evans, J., Fried, L. P., Guralnik, J. M., Katz, P. R., Malmstrom, T. K., McCarter, R. J., Gutierrez Robledo, L. M., Rockwood, K., von Haehling, S., Vandewoude, M. F., and Walston, J. (2013). Frailty Consensus: A Call to Action. Journal of the American Medical Directors Association, 14, 392-397.

Muessig, J. M., Nia, A. M., Masyuk, M., Lauten, A., Sacher, A. L., Brenner, T., Franz, M., Bloos, F., Ebelt, H., Schaller, S. J., Fuest, K., Rabe, C., Dieck, T., Steiner, S., Graf, T., Jánosi, R. A., Meybohm, P., Simon, P., Utzolino, S., … Jung, C. (2018).

Clinical Frailty Scale (CFS) reliably stratifies octogenarians in German ICUs: A multicentre prospective cohort study. BMC Geriatrics, 18(1).

https://doi.org/10.1186/s12877-018-0847-7

Murukesu, R. R., Singh, D. K. A., Shahar, S., & Subramaniam, P. (2020). A Multi-Domain Intervention Protocol for the Potential Reversal of Cognitive Frailty: "WE-RISE" Randomized Controlled Trial. Frontiers in Public Health, 8.

https://doi.org/10.3389/fpubh.2020.00471

Ng, T. P., Feng, L., Nyunt, M. S. Z., Feng, L., Niti, M., Tan, B. Y., Chan, G., Khoo, S. A., Chan, S. M., Yap, P., & Yap, K. B.(2015). Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal among Older Adults: A Randomized Controlled Trial. American Journal of Medicine, 128(11), 1225-1236.e1.

https://doi.org/10.1016/j.amjmed.2015.06.017

National Institute of Health and Care Excellence [NICE]. (2018). Dementia: assessment, management and support for people living with dementia and their carers NICE guideline.

www.nice.org.uk/guidance/ng97

Song, X., Mitnitski, A., & Rockwood, K. (2010). Prevalence and 10-Year outcomes of frailty in older adults in relation to deficit accumulation. Journal of the American Geriatrics Society, 58(4), 681-687.

https://doi.org/10.1111/j.1532-5415.2010.02764.x

Spector, A., Thorgrimsen, L., Woods, B., Royan, L., Davies, S., Butterworth, M., & Orrell, M. (2003). Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: Randomised controlled trial. British Journal of Psychiatry, 183(SEPT.), 248-254.

https://doi.org/10.1192/bjp.183.3.248

Spector, A., Woods, B., Stoner, C. R., & Orrell, M. (2006). Making a difference 1: The manual for group facilitators (1st ed.). Hawker Publications.

Tam, A. C. Y., Chan, A. W. Y., Cheung, D. S. K., Ho, L. Y. W., Tang, A. S. K., Christensen, M., Tse, M. M. Y., & Kwan, R. Y. C. (2022). The effects of interventions to enhance cognitive and physical functions in older people with cognitive frailty: a systematic review and meta-analysis. European Review of Aging and Physical Activity, 19(1).

https://doi.org/10.1186/s11556-022-00299-9

Wallis, S. J., Wall, J., Biram, R. W. S., & Romero-Ortuno, R. (2015). Association of the Clinical Frailty Scale with Hospital Outcomes. Quarterly Journal of Medicine: An International Journal of Medicine, 108(12), 943-949.

ELIGIBILITY:
Stroke Survivors Inclusion Criteria:

* 18+ years old
* Had a stroke 12 months ago, or less
* Due to be discharged back home before the adapted CST group starts
* Experiencing a loss of physical resilience as a result of your stroke
* Experiencing some difficulty with your memory or thinking as a result of your stroke
* Have a family member or friend who regularly supports you and is willing to take part in a connected research study
* Have the ability to speak and read the English language to participate fully in the adapted CST group and online interview

Stroke Survivors Exclusion Criteria:

* Have significant difficulties with language, memory or thinking that would take taking part too difficult
* Are not able to independently make the decision about whether you would like to take part
* Have a diagnosis of dementia
* Do not have access to a computer, laptop or tablet from which you can access an online interview

Carers Inclusion Criteria

* Are 18+ years old
* Regularly support someone who has survived a stroke
* Have the ability to speak and read the English language to engage fully in the CST take-home activities and online interview
* Are able to independently make the decision about whether you would like to take part in the study

Carers Exclusion Criteria

* Do not have access to a computer, laptop or tablet from which you can access an online interview
* Are a professional carer for the person you support
* Are being investigated by the safeguarding team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Stroke Survivors: Stroke Survivors
- Carers: Carers
Period: Overall Study
Arm/Group | Stroke Survivors | Carers
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stroke Survivors | Carers | Total
Number analyzed (Participants) | 5 | 5 | 10
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Educational Level [Count of Participants; unit: Participants]
  O-Level/GCSE | 0 | 2 | 2
  Higher Education | 2 | 2 | 4
  No qualifications | 2 | 0 | 2
  Not disclosed | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Framework Analysis Using the Theoretical Framework of Acceptability as a Guiding Framework
Description: Semi-structured interviews were carried out using a topic guide based on the Theoretical Framework of Acceptability (TFA; Sekhon et al., 2017).
  The resulting data were analysed using Framework Analysis, using the TFA as the guiding framework. The transcripts were coded both deductively and inductively. Deductive codes were based on the definitions of the 7 constructs of the TFA outlined by Sekhon et al. (2017). Any meaningful data relating to acceptability that did not fit within these definitions were inductively coded.
  Because the data for stroke survivors was analysed completely separately from that for carers for the purposes of the researchers producing two independent doctoral theses, the only data that can be compared is that which resulted from the deductive coding. Therefore, the data reported below reports the number of participants who provided meaningful data relating to each of the 7 constructs of the TFA.
Time Frame: 4 weeks
Population: 1 stroke survivor dropped out of intervention mid way through. Both this stroke survivor and their carer were lost to follow-up and did not take part in interviews
Measure: Count of Participants; unit: Participants
Arm/Group | Stroke Survivors | Carers
Number analyzed (Participants) | 4 | 4
Participants
  Affective Attitude - How an individual feels about the intervention | 4 | 4
  Burden - The perceived amount of effort that is required to participate in the intervention | 4 | 4
  Ethicality - The extent to which the intervention had a good fit with an individual's value system | 4 | 4
  Intervention Coherence - The extent to which they understand the intervention and how it works | 4 | 4
  Opportunity Costs - The extent to which benefits or values must be given up for the intervention | 3 | 4
  Perceived Effectiveness - The extent to which the int. is perceived as likely to achieve its purpose | 4 | 4
  Self-Efficacy - The participant's confidence in their ability to participate in the intervention | 4 | 4

ADVERSE EVENTS:
Time Frame: From enrollment until end of interviews, up to 13 weeks
Arm/Group | Stroke Survivors | Carers
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stroke Survivors (N=5) | Carers (N=5)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — existing condition was exacerbated in one carer as a result of supporting the stroke survivor to attend the intervention (pushing wheelchair through hospital)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT06733103/Prot_SAP_000.pdf